CLINICAL TRIAL: NCT01858545
Title: An Evaluation of Tissue Engineering Approaches for Treatment of Neuropathic Diabetic Foot Ulcers Resistant to Standard of Care: A Prospective, Randomized Controlled Trial
Brief Title: A Comparative Efficacy Study: Treatment for Non-healing Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACL2011-002-I
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): MatriStem MicroMatrix and MatriStem Wound Matrix
  Interventions: Device: MatriStem
- Comparator (Active Comparator): Cellular Dermal Replacement Tissue
  Interventions: Device: Cellular Dermal Replacement Tissue

INTERVENTIONS:
Device: MatriStem — MatriStem MicroMatrix and MatriStem Wound Matrix
  Arms: Experimental
Device: Cellular Dermal Replacement Tissue — Cellular Dermal Replacement Tissue
  Arms: Comparator

SUMMARY:
The primary objective of this study is to assess the effectiveness of MatriStem devices compared to cellular dermal replacement tissue, for the treatment of non-healing diabetic foot ulcers.

DETAILED DESCRIPTION:
Due to their characteristically poor healing capacity, diabetic foot ulcers (DFUs) are challenging for clinicians to treat. This prospective, multi-center clinical study will examine outcomes following treatment of DFUs, with one of two FDA cleared tissue-engineered devices, MatriStem® or cellular dermal replacement tissue, on DFUs that have demonstrated an inadequate response to initial standard of care therapy. The incidence of ulcer closure, rate of wound closure, and quality of life will be evaluated over a eight week period.

ELIGIBILITY:
Major Inclusion Criteria:

* Subject has a current diagnosis of type I or type II diabetes
* Subject's ulcer is on the forefoot or heel
* Subject has chronic ulcer - has been present for minimum of 4 weeks
* Subject's ulcer extends through the dermis and into the subcutaneous tissue
* Subject's HgbA1c <12%
* Subject has adequate circulation to the study foot as evidenced by a Doppler measured ABI greater than or equal to 0.7after 10 minutes rest

Major Exclusion Criteria:

* Subject has a known sensitivity to bovine- or porcine-derived products.
* Subject's ulcer is due to a non-diabetic etiology
* Subject's ulcer is over a Charcot deformity of the mid-foot
* Subject's random blood sugar readings are >450 mg/dL
* Subject is on dialysis
* Subject has a non-study ulcer on the study limb located within 7.0 cm of the study ulcer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gilbert, PhD, Study Director — Integra LifeSciences
Locations (9):
- United States (9):
  - Carl t. Hayden Phoenix VA Medical Center, Phoenix, Arizona
  - Associated Foot & Ankle Specialists, PC, Phoenix, Arizona
  - Center for Clinical Research Inc., Castro Valley, California
  - Valley Vascular Surgery Associates, Fresno, California
  - Denver VA Medical Center, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Advanced Research Institute of Miami, Homestead, Florida
  - NewPhase Clinical Trials, Corp., Miami Beach, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Comparator
Started | 27 | 29
Completed | 23 | 23
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Comparator | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (9.8) | 58.5 (11.4) | 57.6 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Wound Closure
Description: Number of participants with incidence of complete wound closure
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Comparator
Number analyzed (Participants) | 27 | 29
Participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | Experimental | Comparator
Serious Adverse Events (participants affected / at risk) | 5/27 | 2/29
Other Adverse Events (participants affected / at risk) | 1/27 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=27) | Comparator (N=29)
Enteritis (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Localized Infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular Accident (Death) (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=27) | Comparator (N=29)
Wound Infection (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes